CLINICAL TRIAL: NCT03290755
Title: Sexual Hepatitis C in HIV Positive Men Who Have Sex With Men (MSM) in Bordeaux
Acronym: HEPCSEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/01
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Human Immunodeficiency Virus (HIV); Hepatitis c
Keywords: Hepatitis C; sexual network; sexual transmitted; men who have sex with men; HIV positive; sexual behaviour
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Homosexuality; HIV Seropositivity; Coitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSM co-infected HIV-HCV
  Interventions: Behavioral: semi-directed interviews

INTERVENTIONS:
Behavioral: semi-directed interviews — semi-directed interviews in order to collect socio-behavioral data

SUMMARY:
The main objective of this study is to analyse sexual behavior of HIV + MSM in Bordeaux, who have sexually contracted hepatitis C between January 1st 2013, to January 31, 2017. These data will bring some improvement about prevention and maybe reduced the hepatitis C incidence.

DETAILED DESCRIPTION:
Hepatitis C (HCV) is considered in part as a sexually transmitted infection (STI). A marked decrease in its incidence has been observed for several years, coinciding with the availability of new direct acting antiviral treatments (DAA). However, people are increasingly infected with the hepatitis C virus, especially HIV-positive MSM. This increase is explained by new sexual practices that are particularly at high level of risk, despite the widening accessibility of new DAA. Prevention also plays an important role in implementing an effective risk reduction policy. New methods of prevention must therefore be developed. For this purpose, it is imperative to know the natural history of acute hepatitis C, the different behaviours at risk of HCV transmission, and the demonstration of socio-sexual networks (clusters) thanks to virological phylogenetic studies. In order to improve hepatitis C prevention, we wish to establish a descriptive study focusing on :

* Descriptive analysis of the natural history of hepatitis C,
* Identification of patient clusters (phylogenetic analysis)
* Description of the sexual behaviors of infected patients, through a semi-directed interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* HIV-1 and/or HIV-2 confirmed Infection
* Men who have sex with Men
* Patients included in the "ANRS CO3Aquitaine cohort".
* HCV contamination documented over the period 01/01/2013 to 01/31/2017 (A positive HCV serology and a HCV plasma RNA positive) AND a negative HCV serology OR a positive HCV serology and a negative plasma RNA before inclusion period
* A person who has received information about the protocol and has given oral consent and that his / her non-opposition is documented in his / her medical file.

Exclusion Criteria:

* Transfusion contamination
* Substance abuse IV out of SLAM context
* Refusal to consent to research.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who have sex with Men co-infected HIV-HCV
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Analyse sexual behaviours among HIV positive MSM in Bordeaux, through semi-directed interviews | At inclusion (day 0)

SECONDARY OUTCOMES:
Identifying socio-sexual networks through phylogenetic analysis | At inclusion (day 0)
Describing the natural history of sexual hepatitis C in HIV positive MSM | At inclusion (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Linda WITTKOP, MD, PhD, Study Chair — Université de Bordeaux - ISPED - Inserm 2129 - CHU de Bordeaux; Charles CAZANAVE, Prof, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service des Maladies Infectieuses et Tropicales, Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No